CLINICAL TRIAL: NCT05224739
Title: Retrospective International Multicenter Study to Validate the Difficulty Scoring System and Develop a Novel Scoring System for Laparoscopic and Robotic Liver Resections
Brief Title: Validate the Difficulty Scoring System and Develop a Novel Scoring System for Laparoscopic and Robotic Liver Resections
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 020.HPB.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent MILR from January 1, 2000 to December 31, 2020: Hospital of patients who underwent MILR from January 1, 2000 to December 31, 2020.
  Interventions: Procedure: Minimally Invasive Liver Resection

INTERVENTIONS:
Procedure: Minimally Invasive Liver Resection — laparoscopic and robotic liver resections

SUMMARY:
To validate the Iwate difficulty scoring system and Institut Mutualiste Montsouris (IMM) scoring system (Appendix 2) in both laparoscopic and robotic liver resections

DETAILED DESCRIPTION:
Minimally-invasive liver resections (MILR) are increasingly conducted world-wide today. Several international consensus meetings were convened to enable the safe dissemination of laparoscopic and robotic liver resections. The Iwate difficulty scoring system (Appendix 1) was formulated in Japan to grade the difficulty of liver resections. This was to allow beginners to adopt a stepwise approach to safely perform MILR according to their experience and competency level. Although this system has been recently validated in a recent Japanese multicenter study, it has not been externally validated in a large cohort of patients. Thus far, it has only been validated in several small single center studies. Furthermore, its utility for robotic liver resections has not been well-studied.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients operated at a single institution during a fixed period
* Most recent operation date allowed (up till December 31, 2020, to allow three months follow-up).
* All minimally invasive hepatectomy approaches can be included, including lap- assisted (hybrid), hand-assisted, robotic-assisted and pure laparoscopy.
* The data of all patients including those that had repeat liver resections, concomitant surgeries (e.g. colectomies, hilar lymph node dissection, enbloc resections) may be included
* Patients with no "liver tumors" such as recurrent pyogenic cholangitis/ gallbladder may be included
* The site of the "lesion/ pathology" will be considered as the tumor site, size will be considered less than 3 cm unless tumor invades the liver.

Exclusion Criteria:

* • Patients < 18 years of age

  * Patients with liver transplant living donor hepatectomies

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital of patients who underwent Minimally Invasive Liver Resection from January 1, 2000 to December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2024-11-16 (Estimated)

PRIMARY OUTCOMES:
Iwate scores for laparoscopic and robotic liver resections | January 1, 2000 to December 31, 2020
  To validate the Iwate difficulty scoring system IMM scoring system in both laparoscopic .and robotic liver resections. The IWATA measures the difficulty index from 0 to 12. The IMM scoring is from code 1 to 11.

SECONDARY OUTCOMES:
Propensity scores for robotic and laparoscopic liver resections | January 1, 2000 to December 31, 2020
  To perform a propensity score matching (including adjustment for difficulty) comparing robotic and laparoscopic liver resections.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, MD, Principal Investigator — Methodist Health System
Locations (1):
- Liver Institute of Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No